CLINICAL TRIAL: NCT03775733
Title: A 12 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate The Efficacy and Safety of Hydrolysed Red Ginseng Extract on Improvement of Hyperglycemia
Brief Title: Efficacy and Safety of Hydrolysed Red Ginseng Extract on Improvement of Hyperglycemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GH-HG-HR
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Hyperglycemia
Keywords: Hydrolysed red ginseng extract; Glucose; Clinical Trial
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrolysed red ginseng extract (Experimental): Hydrolysed red ginseng extract 2.4g/day for 12 weeks
  Interventions: Dietary Supplement: Hydrolysed Red Ginseng Extract
- Placebo (Placebo Comparator): Placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hydrolysed Red Ginseng Extract — Hydrolysed Red Ginseng Extract 2.4g/day for 12 weeks.
  Arms: Hydrolysed red ginseng extract
Dietary Supplement: Placebo — Placebo for 12 weeks.
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of hydrolysed red ginseng extract on improvement of Hyperglycemia.

DETAILED DESCRIPTION:
This study was a 12 weeks, randomized, double-blind, placebo-controlled human trial. Twenty subjects were randomly divided into Hydrolysed Red Ginseng extract or a placebo group. Fasting and postprandial glucose profiles during oral glucose tolerance test (OGTT) were assessed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-80 years with fasting glucose 100-140 mg/dL

Exclusion Criteria:

* Weight less than 48 kg or weight decreased by more than 10% within past 3 months
* Have clinically significant acute or chronic cardiovascular system, endocrine system, immune system, respiratory system, hepatic biliary system, kidney and Urinary system, neuropsychiatry, musculoskeletal, inflammatory and hematologic malignancies, gastrointestinal disorders, etc.
* Hypoglycemic agent, Obesity medicine, Lipid lowering agent within past 3 months
* Blood sugar improvement or healthy functional food within past 1 month
* Under antipsychotic medication therapy within past 2 months
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test by show the following results

  * aspartate aminotransferase, alanine aminotransferase > Reference range 3 times upper limit
  * Serum Creatinine > 2.0 mg/dl
* Pregnancy or breast feeding
* If a woman of childbearing doesn't accept the implementation of appropriate contraception
* Principal Investigator judged inappropriate for participation in study because of Laboratory test result, etc.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-07 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of blood glucose | 12 weeks
  Changes of fasting and postprandial glucose during OGTT were assessed before and after the intervention.

SECONDARY OUTCOMES:
Changes of blood insulin | 12 weeks
  Changes of blood insulin during OGTT were assessed before and after the intervention.
Changes of area under the curve of Glucose and Insulin | 12 weeks
  Changes of area under the curve of Glucose and Insulin were assessed before and after the intervention.
Changes of Homeostatic model assessment-insulin resistance | 12 weeks
  Changes of physiological parameter{Homeostatic model assessment-insulin resistance(mg/dl)} were assessed before and after the intervention.
Changes of Homeostatic model assessment-beta-cell | 12 weeks
  Changes of physiological parameter{Homeostatic model assessment-beta-cell(mg/dl)} were assessed before and after the intervention
Changes of HbA1c | 12 weeks
  Changes of HbA1c(%) were assessed before and after the intervention
Changes of C-peptide | 12 weeks
  Changes of C-peptide(ng/ml) were assessed before and after the intervention.
Changes of lipid profile | 12 weeks
  Changes of lipid profile were assessed before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea